CLINICAL TRIAL: NCT00482443
Title: A Multinational, Randomised Study of the Efficacy of the Diabetes Interactive Diary (DID), a Carbohydrates/Insulin Bolus Calculator and a Telemedicine System Based on the Communication Between Physician or Dietitian and Patient by SMS
Brief Title: Assessing the Effectiveness of Diabetes Interactive Diary (DID) in Diabetes Management
Acronym: DID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Royal Bournemouth Hospital (Other)
Responsible Party: Professor David Kerr., Royal Bournemouth Hospital.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DID
Record Dates: First submitted 2007-06-04; First posted 2007-06-05 (Estimated); Last update posted 2008-07-10 (Estimated); Status verified 2008-07

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): To assess the efficacy of a Diabetes Interactive Diary in Diabetes Management.
  Interventions: Other: A software programme in mobile telephone
- 2 (Active Comparator): Control Arm. Patients will receive standard education programme.
  Interventions: Other: Standard Education Programme.

INTERVENTIONS:
Other: A software programme in mobile telephone — Use of Mobile phone technology in maintaining Diabetes Interactive Diary.
  Arms: 1
Other: Standard Education Programme. — Control Arm patients will receive a standard education programme designed to help the Type 1 Diabetic manage their condition.
  Arms: 2

SUMMARY:
For people with Type 1 Diabetes, blood glucose control is achieved by matching insulin doses directly to the amount of carbohydrate consumed. We are looking at new ways to help our patients with type 1 diabetes manage their diabetes control more effectively. We are testing if "Diabetes Interactive Diary" (DID), a novel programme designed to be used on a mobile phone, can represent an important tool in carbohydrate counting while avoiding the use of complex calculations and in depth knowledge about the carbohydrate content of their food.

DETAILED DESCRIPTION:
This is randomized control trial aimed to evaluate the effectiveness of a DID compare to the standard education approach in order to help the patients with Type 1 diabetes to estimate the carbohydrate in their food and adjust insulin doses. It involves individuals with Type 1 diabetes who are not habitually using carbohydrate counting. They should be testing their blood sugar levels at least 3 times a day, using multiple daily injections of short-acting and long-acting insulin analogues, with HbA1c between 7.5% and 10% and are familiar with the use of mobile phones and possess a personal SIM card.

Patients will be randomized to the standard education programme run for 4 full days over a 4 week period or to the DID programme run as three 2-hour sessions over a two-week period.

The DID is a novel software programme installed on the patient's mobile telephone. It facilitates the communication between the dietitian and the patient by using SMS text messages, so that the dietitian can monitor glycaemic control and suggest adjustments if necessary. It can be described as a little computer, where the patient can record their blood glucose value, the amount of insulin injected and the amount of carbohydrate consumed.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or over
* Not habitually using carbohydrate counting and insulin dose adjustment
* Testing their blood sugar levels at least 3 times a day
* Using multiple daily injections of short-acting and long-acting insulin analogues
* With HbA1c between 7.5% and 10%
* Familiar with the use of mobile phones and possess a personal SIM card.

Exclusion Criteria:

* Mental conditions, depression or high anxiety rendering the subject unable to understand the nature, scope, and possible consequences of the study
* Eating disorders
* Pregnancy
* Any clinically significant major organ system disease or infective diseases
* Any disease or condition or abuse of illicit drugs, prescription medicines or alcohol that in the opinion of the investigator may interfere with the completion of the study
* Subject unlikely to comply with protocol, e.g., uncooperative attitude, inability to return for follow-up visits and unlikely to complete the study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-03; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
The difference in HbA1c between the patient in the DID group and in the standard education group. | 6 month

SECONDARY OUTCOMES:
The differences between the two groups in terms of, lipid profile, blood pressure, the number of hypoglycaemic episodes, daily blood sugar fluctuation, total insulin dose, weight changes and patients' satisfaction with the treatment. | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: David Kerr, Doctor, Principal Investigator — Royal Bournemouth Hospital; Anita Bowes, Dietitian, Principal Investigator — Royal Bournemouth Hospital
Locations (1):
- Royal Bournemouth Hospital, Bournemouth, Dorset, United Kingdom